CLINICAL TRIAL: NCT05523310
Title: Prospective, Observational Study to Assess Migraine Prediction Tool Based on Prodromal Symptoms and Additional Parameters
Brief Title: Observational Study to Assess Migraine Prediction Tool
Status: Suspended | Type: Observational
Why Stopped: The Sponsor decided to cancel the study due to commercial considerations
Sponsor: Theranica (Industry)
Responsible Party: Sponsor
Other Study IDs: TCH010
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-10

CONDITIONS: Migraine
Keywords: Migraine prediction; Migraine prodrome; Migraine prevention
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Training group: The training group will be used to develop the prediction model, based on their reported daily questionnaire. Participants in the training group will not be included in the Validation group
  Interventions: Other: Daily questionnaire
- Validation group: The validation group will be used only for validation (test) of the prediction model ("Naïve group"). Participants in the validation group could not be recruited from the training group
  Interventions: Other: Daily questionnaire

INTERVENTIONS:
Other: Daily questionnaire — All patients will be asked to complete a daily questionnaire regarding their migraine, medications, and prodromal symptoms during that day

SUMMARY:
This is a prospective, observational study. The participant will be required to approve his/her participation in the study by completing the electronic consent form. Data collected within the first eight weeks (weeks 1-8) will be used to develop the prediction models (either personal or population/group models). The developed algorithm will be freezer and tested against the data collected during weeks 1-8 of a different cohort population

DETAILED DESCRIPTION:
Migraine treatment may be acute (abortive) or preventive (prophylactic), with patients often requiring both. The objectives of acute treatment are to treat attacks early; to achieve quick pain relief; to minimize or eliminate adverse events; to restore function; to decrease recurrence and the need for rescue treatment; and to reduce medical resource use. Preventive treatment is aimed to lower the frequency, intensity, and duration of the attacks.

In general, a prodrome is an early sign or symptom (or set of signs and symptoms) that often indicates the onset of a disease before more diagnostically specific signs and symptoms develop. Prodromal or premonitory symptoms occur in about 60% of those with migraines, with an onset that can range from two hours to two days before the start of pain or the aura. These symptoms may include a wide variety of phenomena including altered mood, irritability, depression or euphoria, fatigue, craving for certain food(s), stiff muscles (especially in the neck), constipation or diarrhea, and sensitivity to smells or noise. This may occur in those with either migraine with aura or migraine without aura. Neuroimaging indicates the limbic system and hypothalamus as the origin of prodromal symptoms in migraine.

Robust prediction of migraine attacks could lead to pre-emptive treatment, provide patients with opportunities to plan for impending attacks, reduce interictal anxiety, and improve self-efficacy among other benefits.

This study aims to develop and evaluate the effectiveness of a migraine prediction tool based on early prodromal (pre-migraine) symptoms, that may enhance the acute treatment of migraine

Prior enrollment, Informed consent must be obtained from each participant before any protocol-related activities are performed. Participants will receive a daily notification (through an app notification) with a link to the daily questionnaire. The app may collect other data items, related to the specific location of every participant, such as weather, air quality, etc.

The primary outcome measure is the presence of headache attack occurring over the 24-hour period recorded following a daily diary entry.

During the development phase, 100% of the data will be used for developing and training the prediction model. Once the model will be ready, it will be "freezer" and used over a different cohort population to validate the prediction model. The AUC of the prediction model will be assessed to validate the accuracy (Specificity vs. Sensitivity) of the prediction model.

The study will include the development of a general predictive model for the study population, with adjustments to individual participants, forecasting the probability of experiencing a headache and/or aura phase of a migraine attack during a particular interval. The outcome measure performance of this model using the Area Under the Curve (AUC) metric. The AUC model measures how often the algorithm predicts a higher probability for a migraine over non-migraine.

ELIGIBILITY:
I

Inclusion Criteria:

* Subject age 18-75 years.
* Subject has migraine diagnosis for over 6 months prior to enrolling to the study.
* Subject has 4-24 headache days per month.
* Subject has a Nerivio user account, or willing to create a Nerivio user account to participate in the study.
* Subject is willing to sign an Informed Consent Form.

Exclusion Criteria:

• NA

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population consists of migraineurs who have already used Nerivio and its mobile application prior to joining the study and those who have not, with a target ratio of 50:50 (and up to 30:70 or 70:30) between these two subject types
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2030-01-01 (Estimated); Primary Completion 2030-10-01 (Estimated); Study Completion 2030-11-15 (Estimated)

PRIMARY OUTCOMES:
Validation of an effective algorithm and software to predict migraine attacks. | Predication period of 24 hours prior headache
  The primary endpoint will be the Predivio's prediction model sensitivity and specificity, presented by receiver operating characteristic (ROC) analysis using the Area Under the Curve (AUC) within the validation cohort population

SECONDARY OUTCOMES:
Predivio accuracy | Predication period of 24 hours prior headache
  Predivio's accuracy will be evaluated by the sensitivity and specificity, presented by the Area Under the Curve (AUC) within the validation cohort population
Predivio's percent of participants for whom the sensitivity and specificity are at least 80%. | Predication period of 24 hours prior headache
  Predivio's percent of participants will be evaluated by the sensitivity and specificity of at least 80% within the validation cohort population

OTHER OUTCOMES:
Difference in prescribed medications usage | 8 weeks
  The difference in the usage of prescribed medications for acute treatment of migraine between subjects using Nerivio as an acute therapy and those who do not. The average number of "migraine medication days" throughout the study will be compared between the groups.
Health economics analysis | 8 weeks
  Health economics analysis of the difference between subjects using Nerivio as a therapy and those who do not with respect to:
  1. Absenteeism - number of missed work/school days
  2. Presenteeism - number of work/school days with moderate/severe functional disability
  3. Healthcare provider appointments
  4. ED visits
  5. Brain MRI/CT scans

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Westport Headache Institute, Westport, Connecticut
  - Headache Neurology Research Institute, Ridgeland, Mississippi
  - Nuvance Health Vassar Medical Center, Poughkeepsie, New York

IPD SHARING:
Plan to Share IPD: No